CLINICAL TRIAL: NCT03497247
Title: Mindfulness-Based Cognitive-Behavioral Therapy for Gambling Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-TCC-2017-102
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive-Behavioral Therapy (Experimental)
  Interventions: Behavioral: Mindfulness-Based Cognitive-Behavioral Therapy
- Cognitive-Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Cognitive-Behavioral Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive-Behavioral Therapy — Both arms have the same intervention techniques (relative intervention, stimulus control and others) except relapse prevention sessions. In the experimental arm, these sessions are carried out from Mindfulness, and in the active comparator is the usual relapse prevention.

SUMMARY:
To compare two group psychological interventions for Gambling Disorder in terms of effectiveness and efficacy. One group is based in cognitive-behavioral therapy (TAU) and the other group is based in TAU with Mindfulness-Based Relapse Prevention (Chawla, Marlatt & Gordon, 2011). Both interventions are composed by 14 weekly sessions, and follow-up to a month, three months, six months, one and two years.

ELIGIBILITY:
Inclusion Criteria:

* Gambling Disorder (DSM-5; APA, 2013).
* 18 years or older.
* Males and females.

Exclusion Criteria:

* Current psychosis or other severe/acute mental disorder.
* Current substance abuse.
* Intellectual disability.
* Under 18 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-06-29 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
South Oaks Gambling Screen (SOGS; Lesieur and Blume, 1987) | 5 minuts
DSM-IV-TR (APA 2000) | 5 minuts
Difficulties in Emotion Regulation Scale (DERS, Gratz and Roemer, 2004) | 5 minuts
Five Facets Mindfulness Questionnaire (FFMQ; Baer et al. 2006) | 5 minuts
EQ-Decentering (Soler et al., 2014) | 5 minuts
Gambling Related Cognitions Scale (GRCS; Raylu & Oei, 2004) | 5 minuts
MBRP - Adherence and Competence Scale (Chawla et al. 2010 | 90 minuts (by co-therapist)

SECONDARY OUTCOMES:
Temperament and Character Inventory-Revised (TCI-R; Cloninger 1999) | 20 minuts
Symptom Checklist-Revised (SCL-90-R; Derogatis 1990) | 20 minuts
UPPS (Whiteside and Lynam, 2001) | 10 minuts
URICA - problem gambling (Gómez-Peña et al. 2011) | 10 minuts
AUDIT (OMS, 1989) | 5 minuts
DUDIT (Berman et al. 2003) | 5 minuts

CONTACTS AND LOCATIONS:
Overall Officials: Marta Sancho, PhD, Principal Investigator — Fundació de Gestió Sanitària de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Santa Creu i Sant Pau Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided